CLINICAL TRIAL: NCT07109908
Title: The Effect of Wiping, Showering and Wrapping Bath Used During the First Bath on Stress Level, Skin Moisture and Physiological Parameters in Neonates Hospitalized in the Neonatal Intensive Care Unit
Brief Title: Stress Level, Skin Moisture and Physiological Parameters in the First Bath of Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Demet Guney, MSc., Research Assist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Kastamonu Unıversity
Record Dates: First submitted 2025-06-30; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Infant Behavior
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wiping Bath (Experimental): The babies in this group were given the first bath in the form of wiping baths. The bathing application was carried out by the midwife working in the unit and experienced in bathing newborns.
  The newborn's clothes except the diaper are removed, the newborn is wrapped in a towel, the newborn's face and body are wiped clean with a skin cleanser and cotton cloth compatible with the baby's skin, the diaper is removed and the genital area is wiped, the baby's body is wiped with a cloth moistened with water (37-39 oc), the body is dried, the baby's body is wrapped in a dry towel, the baby's head is washed with a shampoo compatible with the baby's skin, the baby's head is dried and a hat is put on, The newborn was dressed in clothes.
  Interventions: Behavioral: Wiping Bath
- Wrapping Bath (Experimental): The first bath of the babies in this group was in the form of a wrap-up bath, in which the baby was wrapped and placed in the bathtub. The bathing application was carried out by the midwife working in the unit and experienced in bathing newborns.
  The newborn's clothes were removed, the newborn was wrapped in a towel, the newborn was slowly immersed in water wrapped in a towel in a bathtub with a maximum of 7 cm of water at the appropriate temperature (37-39 oC), the towel was gently opened and the baby's body was gently cleaned with a suitable cleansing product and a cotton swab, including the torso, legs and genital area, the baby's head was wetted and washed with a shampoo compatible with the baby's skin, the baby's head was rinsed by pouring water from the hairline, The baby's torso was gently removed from the bathtub and rinsed, the newborn baby was dried and then dressed in clothes.
  Interventions: Behavioral: Wrapping Bath
- Showering Bath (Experimental): The first bath of the babies in this group was in the form of a shower bath. The bathing application was carried out by the midwife working in the unit and experienced in bathing newborns.
  The newborn's clothes are removed, the newborn's body is soaked with water at the appropriate temperature (37-39 oC) under running water, the body is washed with the appropriate skin cleanser and cotton cloth, the head is washed with the appropriate shampoo for the baby's skin, the whole body is rinsed under running water, the whole body is dried with a towel and the clothes are dressed.
  Interventions: Behavioral: Showering Bath

INTERVENTIONS:
Behavioral: Wiping Bath — The babies in this group were given the first bath in the form of wiping baths. The bathing application was carried out by the midwife working in the unit and experienced in bathing newborns.
  The newborn's clothes except the diaper are removed, the newborn is wrapped in a towel, the newborn's face and body are wiped clean with a skin cleanser and cotton cloth compatible with the baby's skin, the diaper is removed and the genital area is wiped, the baby's body is wiped with a cloth moistened with water (37-39 oc), the body is dried, the baby's body is wrapped in a dry towel, the baby's head is washed with a shampoo compatible with the baby's skin, the baby's head is dried and a hat is put on, The newborn was dressed in clothes.
  Arms: Wiping Bath
Behavioral: Wrapping Bath — The first bath of the babies in this group was in the form of a wrap-up bath, in which the baby was wrapped and placed in the bathtub. The bathing application was carried out by the midwife working in the unit and experienced in bathing newborns.
  The newborn's clothes were removed, the newborn was wrapped in a towel, the newborn was slowly immersed in water wrapped in a towel in a bathtub with a maximum of 7 cm of water at the appropriate temperature (37-39 oC), the towel was gently opened and the baby's body was gently cleaned with a suitable cleansing product and a cotton swab, including the torso, legs and genital area, the baby's head was wetted and washed with a shampoo compatible with the baby's skin, the baby's head was rinsed by pouring water from the hairline, The baby's torso was gently removed from the bathtub and rinsed, the newborn baby was dried and then dressed in clothes.
  Arms: Wrapping Bath
Behavioral: Showering Bath — The first bath of the babies in this group was in the form of a shower bath. The bathing application was carried out by the midwife working in the unit and experienced in bathing newborns.
  The newborn's clothes are removed, the newborn's body is soaked with water at the appropriate temperature (37-39 oC) under running water, the body is washed with the appropriate skin cleanser and cotton cloth, the head is washed with the appropriate shampoo for the baby's skin, the whole body is rinsed under running water, the whole body is dried with a towel and the clothes are dressed.
  Arms: Showering Bath

SUMMARY:
Objectıve: The aim of this study was to determine the effect of wipe (WG), shower (SG) and tub bath (TG) on stress level, skin moisture and physiological parameters used during the first bath in newborns hospitalized in the Neonatal Intensive Care Unit (NICU).

Hypotheses of the Research

Hypothesis 01,2,3: There is no difference between wiping baths, wrapping baths and shower baths in terms of their effects on thermoregulation, stress level, skin moisture and physiological parameters of newborns.

Hypothesis 11: Newborns who are given a wrap-up bath have a lower stress level than if they are swept and showered.

Hypothesis 12: Newborns who are given a wrap-up bath have better skin moisture levels than newborns who are wiped and showered.

Hypothesis 13: Physiological parameters (body temperature, heart peak, respiratory rate, oxygen saturation) of newborns who are given a wrap bath are less affected than wiping and showering.

DETAILED DESCRIPTION:
Bathing in newborns is an important midwifery/nursing practice that not only cleans the baby's skin, but also relaxes the baby (Tambunan and Mediani, 2019; da Fonseca Filho et al., 2017), supports immune system development (Burdall et al., 2019), and contributes to the preservation of skin integrity (Lima et al., 2020). If the appropriate method is not chosen in bathing in newborns and the bath is not performed under appropriate conditions, it may adversely affect the adaptation of the newborn to the extrauterine environment, physiological parameters and stress level. Therefore; the bath should be applied in a warm environment, in a safe and peaceful way, and with the appropriate method (Lima et al., 2020). In addition to performing bathing in the appropriate way, midwives/nurses should take appropriate precautions by observing the physiological parameters and stress responses of infants (Huang et al., 2022; Tambunan et al., 2022).

In newborns, wrap-around bath, wipe bath and shower bath methods are frequently used. Wiping bath is the process of wiping the baby's skin. The wrap-around bathtub bath method is to clean the baby by wrapping it with a soft towel or blanket and placing it in a bathtub filled with water at the appropriate temperature, preserving the flexion and midline position. A bath in the form of a shower is the process of bathing the newborn under running water (Ceylan and Bolışık, 2022; Karakul and Dogan, 2020).

ELIGIBILITY:
Inclusion Criteria:

* Birth weight of 2500 g or more
* Body temperature within the normal range (36-37.3°C)
* Respiratory rate between 30-60 breaths per minute
* Oxygen saturation above 85%
* Absence of neurological problems (e.g., hypotonia, hypertonia)
* Absence of congenital defects
* No dermatological problems
* Parental consent and voluntary participation in the research

Exclusion Criteria:

* Presence of respiratory failure or distress
* Requirement for ventilator support
* Continuous need for high-concentration oxygen via methods such as hood or CPAP
* History of convulsions
* Clinical evidence of infection

Ages: 1 Month to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Physiological Variables Follow-up Form | Just before bathing, just after bathing, and 30 minutes after bathing
  Developed by researchers based on the literature (Taşdemir, 2017; Tibik and Şener, 2024) this form, physiological variables of the newborn; heart rate (min), respiratory rate (min), oxygen saturation value (%SpO2%), body temperature (°C) and neonatal skin condition score were used to record the evaluation results. The physiological parameters of the newborn were evaluated three times in each group: just before, immediately after bathing and 30 minutes after bathing.
Skin Moisture Tracking Form | 6th hour, 12th hour and 24th hour just before and after bath
  Developed by researchers based on the literature (Çeçen, 2023; Taşdemir and Efe, 2025). Skin moisture monitoring was measured with a skin moisture meter and recorded in the form. Skin moisture measurement was made by the same nurse from the determined areas (forehead, abdomen, forearm and upper leg) just before the bath and at the 6th, 12th hour and 24th hour after the bath. The Skin Moisture Meter is used to measure the amount of moisture at any point of the body only by contact with the skin, with its precise measurement feature. The humidity measurement of the device is in the range of 0% - 99.9%. The moisture meter weighs 40° and works effectively at ambient temperatures between 5° and 40° C (Konar et al., 2020).
Neonatal Stress Scale | 10 min before bathing, during bathing, just after bathing, 15 and 30 min after bathing
  The neonatal stress scale was developed by Ceylan and Bolışık (2017) to assess the stress level in premature babies. The scale includes 8 subgroups including facial expression, body color, respiration, activity level, consolation, muscle tone, extremities and posture and consists of a total of 24 items in 3-point Likert type. In scoring, each subgroup is evaluated between 0-2 points. The score obtained from the scale is a minimum of 0 points and a maximum of 16 points. An increase in the score indicates that the baby's stress level has increased. Cronbach's Alpha values of the scale ranged from 0.65 to 0.81 for Observer 1 and 0.69 to 0.78 for Observer 2 (Ceylan and Bolışık 2017). The stress level of the newborns was evaluated 5 times through the Neonatal Stress Scale, 10 minutes before bathing, during the bath, immediately after the bath, 15 minutes after the bath, and 30 minutes after the bath.

CONTACTS AND LOCATIONS:
Overall Officials: demet güney, MSc., Principal Investigator — https://sbf.kastamonu.edu.tr/index.php/boeluemler/ebelik
Locations (1):
- Demet Güney, Kastamonu, Turkey (Türkiye)

REFERENCES:
- [Background] Burdall O, Willgress L, Goad N. Neonatal skin care: Developments in care to maintain neonatal barrier function and prevention of diaper dermatitis. Pediatr Dermatol. 2019 Jan;36(1):31-35. doi: 10.1111/pde.13714. Epub 2018 Dec 2. PMID 30506880
- [Background] Cinar N, Yalnizoglu Caka S, Uslu Yuvaci H. Effect of newborn bathing training with the swaddled and tub bathing methods given to primiparous pregnant women on the mother's experience, satisfaction and newborn's stress during the first bathing of the newborn at home: A mixed method study. Jpn J Nurs Sci. 2020 Oct;17(4):e12363. doi: 10.1111/jjns.12363. Epub 2020 Aug 25. PMID 32844590
- [Background] de Freitas P, Bueno M, Holditch-Davis D, Santos HP, Kimura AF. Biobehavioral Responses of Preterm Infants to Conventional and Swaddled Tub Baths: A Randomized Crossover Trial. J Perinat Neonatal Nurs. 2018 Oct/Dec;32(4):358-365. doi: 10.1097/JPN.0000000000000336. PMID 29782435
- [Background] Edraki M, Paran M, Montaseri S, Razavi Nejad M, Montaseri Z. Comparing the effects of swaddled and conventional bathing methods on body temperature and crying duration in premature infants: a randomized clinical trial. J Caring Sci. 2014 Jun 1;3(2):83-91. doi: 10.5681/jcs.2014.009. eCollection 2014 Jun. PMID 25276751
- [Background] Fernandez D, Antolin-Rodriguez R. Bathing a Premature Infant in the Intensive Care Unit: A Systematic Review. J Pediatr Nurs. 2018 Sep-Oct;42:e52-e57. doi: 10.1016/j.pedn.2018.05.002. Epub 2018 May 18. PMID 29779763
- [Background] Higuchi S, Yoshida S, Minematsu T, Hatano Y, Notsu A, Ichinose T. Comparison of the Effects of Bathing and the Dry Technique on the Skin Condition of Early Neonates: A Prospective Observational Study. Ann Dermatol. 2023 Aug;35(4):256-265. doi: 10.5021/ad.22.098. PMID 37550226
- [Background] Konar MC, Islam K, Roy A, Ghosh T. Effect of Virgin Coconut Oil Application on the Skin of Preterm Newborns: A Randomized Controlled Trial. J Trop Pediatr. 2020 Apr 1;66(2):129-135. doi: 10.1093/tropej/fmz041. PMID 31257430